CLINICAL TRIAL: NCT01232842
Title: Assessment of Stem Cell Heterogeneity in AML in Co-Culture Systems Using X Chromosome Inactivation Patterns
Brief Title: Biomarker Study in Tissue Samples From Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML11B4; COG-AAML11B4 (Other: Children's Oncology Group); NCI-2011-02843 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AAML11B4 (Other: Children's Oncology Group)
Record Dates: First submitted 2010-10-30; First posted 2010-11-02 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia; childhood acute myeloid leukemia/other myeloid malignancies
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Cytogenetic Analysis; Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: cytogenetic analysis
Other: HUMARA assay
Other: fluorescence activated cell sorting
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in tissue samples from patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the frequency of acute myeloid leukemia (AML) that originates in CD33+ precursors or in which uncontrolled growth is restricted to CD33+ precursors.

OUTLINE: Cryopreserved acute myeloid leukemia cell samples are separated from endothelial cell by fluorescent-activated cell sorting (FACS) and analyzed for X-chromosome inactivation patterns by cytogenetic/molecular analysis and/or Humara assay.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with acute myeloid leukemia
* Known CD34+ progenitor cells
* Available freshly isolated, uncultured cell samples

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosed with acute myeloid leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-10; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Frequency of AML that originate in CD33+ or in which uncontrolled growth is restricted to CD33+ precursors
Extent of clonal hematopoiesis in small numbers of AML cells

CONTACTS AND LOCATIONS:
Overall Officials: Roland Walter, MD, PhD, Principal Investigator — Fred Hutchinson Cancer Center